CLINICAL TRIAL: NCT06639490
Title: Efficacy of RUS GA Surgical Navigation for Robot-assisted Distal Gastrectomy in Gastric Cancer Patients: Global Multicenter Randomized Controlled Trial
Brief Title: Efficacy of RUS GA Surgical Navigation for Robot-assisted Distal Gastrectomy in Gastric Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1-2024-0044
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group A (Experimental): Robot-assisted gastrectomy will be performed using RUS GA
  Interventions: Device: RUS GA
- Active Comparator Group B (standard treatment) (Active Comparator): Robot-assisted gastrectomy will be performed using without software RUS GA. Only
  Interventions: Procedure: standard treatment

INTERVENTIONS:
Device: RUS GA — he RUS GA (Endoscopic Imaging Treatment Planning Software, E04010.01(2)) is an endoscopic imaging treatment planning software program. It creates a patient-specific simulation of the actual intra-abdominal surgical environment, allowing for the visualization of vascular structures and intra-abdominal organs during the surgical planning process and the operation. RUS GA utilizes preoperative CT images of the patient to segment organs and blood vessels and reconstructs them into a 3D model. Although there is no direct intervention with the patient, the surgeon uses RUS GA as a surgical navigation tool to simulate the surgery before performing the actual procedure.
  Arms: Experimental Group A
Procedure: standard treatment — Only standard treatment is performed.(Robot-assisted gastrectomy will be performed using without software RUS GA.)
  Arms: Active Comparator Group B (standard treatment)

SUMMARY:
This investigator-initiated, randomized superiority clinical trial aims to demonstrate the clinical effectiveness of RUS GA Surgical Navigation, an endoscopic imaging treatment planning software, in patients undergoing robotic-assisted distal gastric cancer surgery. The trial will compare the experimental group using RUS GA with a control group, aiming to show an 8.7% reduction in total surgery duration. The study will involve global multicenter patient recruitment and evaluate the clinical safety and feasibility of the software, which has been shown to be reliable in previous studies.

* Investigational Medical Device: RUS GA (Endoscopic Imaging Treatment Planning Software, E04010.01)
* Clinical Trial duration: 30 months from IRB approval -Target number of subjects: Total of 330 participants

DETAILED DESCRIPTION:
After selecting subjects and obtaining informed consent, randomization will be conducted. Robot-assisted gastrectomy will be performed using RUS GA or without software. Clinical significance will be evaluated through outpatient follow -ups for up to one month after discharge.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals diagnosed with gastric cancer and scheduled for robot-assisted gastrectomy.
2. Adults aged 20 and above who are capable of independent judgment.
3. Individuals capable of undergoing CT imaging according to the prescribed protocol.
4. Individuals who, before participating in the clinical trial, undergo an interview in a separate place, understand sufficient explanation of the purpose and content of the trial, and voluntarily sign informed consent form (approved by the Institutional Review Board)

Exclusion Criteria:

1. Vulnerable individuals (those lacking decision-making capacity, illiterate individuals, pregnant women, newborns, minors under the age of 20, etc.).
2. Patients who cannot undergo CT imaging according to the prescribed protocol before gastric cancer surgery (due to contrast agent allergies, creatinine levels exceeding 1.5 times the normal upper limit, claustrophobia, etc.).
3. Individuals whose major gastric or intra-abdominal arterial/venous structures have been altered due to previous gastric or other abdominal surgeries (however, those with a history of intra-abdominal surgery that did not affect the stomach or major blood vessels are eligible).
4. Patients with a history of residual gastric cancer from previous surgery.
5. Patients who do not consent to participate in the study or withdraw their consent.
6. Patients scheduled for simultaneous resection of other organs besides the stomach.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2024-12-03 (Actual); Primary Completion 2027-02-20 (Estimated); Study Completion 2027-03-22 (Estimated)

PRIMARY OUTCOMES:
Surgery duration | during surgery(Record anesthesia time, total operation time, and robot console time separately)
  To assess whether the use of the endoscopic imaging treatment planning software, RUS GA, in actual surgeries of patients with gastric cancer results in a statistically significant reduction in total surgical time compared to surgeries conducted without the use of RUS GA.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided